CLINICAL TRIAL: NCT04359355
Title: Development and Validation of a New Artificial Intelligence System for Automated Detection of Colorectal Polyps During Colonoscopy
Brief Title: Computer-aided Detection of Colorectal Polyps
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Timo Rath, Professor of Endoscopy, University of Erlangen-Nürnberg Medical School
Other Study IDs: CAID
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Adenoma Colon; Polyp of Colon
Keywords: colonoscopy; endoscopy; adenoma detection; polyp detection; artificial intelligence
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Artificial Intelligence
  Interventions: Device: Artificial Intelligence System for Detection of colorectal polyps

INTERVENTIONS:
Device: Artificial Intelligence System for Detection of colorectal polyps — In this group, an artificial Intelligence System will be used for computer-aided diagnosis of colorectal polyps. Diagnostic Performance of the artificial intelligence System for detection of polyps will be compared against Operator-based detection in the same group

SUMMARY:
In this observational pilot study, we assess the diagnostic performance of an artificial intelligence sytem for automated detection of colorectal polyps.

DETAILED DESCRIPTION:
During standard colonoscopy, a substantial number of colorectal polyps can be missend. As shown in a recent meta-analysis, miss rates for adenomas can reach up to 26%. In this study, it is tested whether an artificial intelligence system that highlights colorectal polyps during screening or surveillance colonoscopy in real time can lead to an increased detection of colorectal polyps during the examination.

ELIGIBILITY:
Inclusion Criteria:

* Screening or surveillance colonoscopy

Exclusion Criteria:

* known or suspected inflammatory bowel disease
* uncontrolled coagulopathy
* known polyps or referral for polypectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting between January and May 2020 for surveillance or Screening colonoscopy in the Ludwig Demling Endoscopy Center of Excellence will be prospectively included under the above mentioned inclusion and exclusion criteria. Prior to enrollment, written informed consent will be obtained.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility to use the AI System in vivo during colonoscopy | 4 month
  As a Primary outcome, whether the AI System is capable of detecting colorectal polyps in vivo during colonoscopy

SECONDARY OUTCOMES:
Diagnostic Performance of the AI System for detecting colorectal polyps | 4 month
  As a secondary outcome, we assess the diagnostic Performance of the AI System for detecing colorectal Polyp in real time

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No
The study will be published in scientific magazines after competion and thus will be made available to other Researchers. Individual Patient data will not be displayed or shared.

REFERENCES:
- [Derived] Pfeifer L, Neufert C, Leppkes M, Waldner MJ, Hafner M, Beyer A, Hoffman A, Siersema PD, Neurath MF, Rath T. Computer-aided detection of colorectal polyps using a newly generated deep convolutional neural network: from development to first clinical experience. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e662-e669. doi: 10.1097/MEG.0000000000002209. PMID 34034272